CLINICAL TRIAL: NCT00290264
Title: A Comparison of Symbicort Single Inhaler Therapy (Symbicort Turbohaler 160/4.5 μg, 1 Inhalation b.i.d. Plus as Needed) and Conventional Best Practice for the Treatment of Persistent Asthma in Adolescents and Adults - a 26-week, Randomised, Open-label, Parallel-group, Multi-centre Study (SALTO)
Brief Title: SALTO - Symbicort Single Inhaler Therapy Use in Adolescent Adults and Adults With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5890L00009; Eudract No: 2004-001107-36; SALTO
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide, Formoterol Fumarate Drug Combination

INTERVENTIONS:
Drug: Budesonide/formoterol
  Other Names: Symbicort

SUMMARY:
The primary objective is to compare the efficacy of Symbicort Single inhaler Therapy with treatment according to conventional best practice in adolescent and adult patients with persistent asthma.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of 3 months documented history of asthma, diagnosed according to the American Thoracic Society (ATS) definition.
* Prescribed inhaled GCS at a dose of ≥320 µg/day and within the approved label for the relevant drug during the last 3 months prior to Visit 1.

Exclusion Criteria:

* Use of any b-blocking agent, including eye-drops.
* Use of oral GCS as maintenance treatment.
* Known or suspected hypersensitivity to study therapy or excipients.
* A history of smoking ≥ 10 pack years (1 pack year = 1 pack (20 cigarettes) per day for one year or equivalent).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2004-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Time to first severe asthma exacerbation

SECONDARY OUTCOMES:
Number of severe asthma exacerbations
Mean use of as-needed medication
Prescribed asthma medication
Peak Expiratory Flow (PEF)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Belgium Medical Director, MD, Study Director — AstraZeneca
Locations (209):
- Belgium (205):
  - Research Site, Aalst
  - Research Site, Aartrijke
  - Research Site, Alsemberg
  - Research Site, Anderlecht
  - Research Site, Angleur
  - Research Site, Ans
  - Research Site, Antwerp
  - Research Site, Anzegem
  - Research Site, Arlon
  - Research Site, Asse
  - Research Site, Aywaille
  - Research Site, Balen
  - Research Site, Barry
  - Research Site, Bastogne
  - Research Site, Battice
  - Research Site, Bellaire
  - Research Site, Berchem
  - Research Site, Bertrix
  - Research Site, Beyne-Heusay
  - Research Site, Bilzen
  - Research Site, Binche
  - Research Site, Bois-de-Villers
  - Research Site, Bornem
  - Research Site, Bouillon
  - Research Site, Boussu
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Burdinne
  - Research Site, Casteau
  - Research Site, Champion
  - Research Site, Chapelle-lez-Herlaimont
  - Research Site, Charleroi
  - Research Site, Châtelet
  - Research Site, Chênée
  - Research Site, Corbion
  - Research Site, Couillet
  - Research Site, De Pinte
  - Research Site, Dendermonde
  - Research Site, Deurne
  - Research Site, Diksmuide
  - Research Site, Dinant
  - Research Site, Dour
  - Research Site, Durnal
  - Research Site, Dworp
  - Research Site, Ekeren
  - Research Site, Elversele
  - Research Site, Erembodegem
  - Research Site, Erquelinnes
  - Research Site, Escanaffles
  - Research Site, Essen
  - Research Site, Etterbeek
  - Research Site, Evere
  - Research Site, Evergem
  - Research Site, Écaussinnes-d'Enghien
  - Research Site, Fleurus
  - Research Site, Frameries
  - Research Site, Ganshoren
  - Research Site, Geluwe
  - Research Site, Genk
  - Research Site, Geraardsbergen
  - Research Site, Ghent
  - Research Site, Gilly
  - Research Site, Godinne
  - Research Site, Gozée
  - Research Site, Grand-Halleux
  - Research Site, Graty
  - Research Site, Grivegnée
  - Research Site, Ham-sur-Heure
  - Research Site, Hamme
  - Research Site, Hannut
  - Research Site, Harzé
  - Research Site, Hasselt
  - Research Site, Havinnes
  - Research Site, Havré
  - Research Site, Heist-op-den-Berg
  - Research Site, Heppen
  - Research Site, Herent
  - Research Site, Herentals
  - Research Site, Herk-de-Stad
  - Research Site, HermalleSousArgenteau
  - Research Site, Herstal
  - Research Site, Hever
  - Research Site, Hoeselt
  - Research Site, Hooglede
  - Research Site, Hornu
  - Research Site, Houthalen-Helchteren
  - Research Site, Huldenberg
  - Research Site, Ieper
  - Research Site, Ingelmunster
  - Research Site, Izegem
  - Research Site, Kalmthout
  - Research Site, Kinrooi-Ophoven
  - Research Site, Kobbegem
  - Research Site, Koksijde
  - Research Site, Kontich
  - Research Site, Koolskamp
  - Research Site, Kortrijk
  - Research Site, Kraainem
  - Research Site, Lauwe
  - Research Site, Leignon
  - Research Site, Leuven
  - Research Site, Libin
  - Research Site, Libramont-Chevigny
  - Research site, Lier
  - Research Site, Liège
  - Research Site, Lobbes
  - Research Site, Lokeren
  - Research Site, Lommel
  - Research Site, Louveigné
  - Research site, Lustin
  - Research Site, Maasmechelen
  - Research Site, Malmedy
  - Research Site, Manage
  - Research Site, Marche-en-Famenne
  - Research Site, Marchovelette
  - Research Site, Massemen
  - Research Site, Mechelen
  - Research Site, Meix-devant-Virton
  - Research Site, Menen
  - Research Site, Merbes-le-Château
  - Research site, Merksem
  - Research Site, Messancy
  - Research site, Mettet
  - Research Site, Middelkerke
  - Research Site, Moerkerke
  - Research Site, Mol
  - Research Site, Monceau-sur-Sambre
  - Research Site, Mons
  - Research site, Mont-Gauthier
  - Research Site, Mont-sur-Marchienne
  - Research Site, Montegnée
  - Research site, Montigny-le-Tilleul
  - Research Site, Moorsel
  - Research Site, Mortier
  - Research Site, Mouscron
  - Research Site, Munkzwalm
  - Research Site, Munsterbilzen
  - Research Site, Musson
  - Research Site, Namur
  - Research Site, Natoye
  - Research Site, Nieuwenrode
  - Research Site, Nieuwkerke
  - Research Site, Nivelles
  - Research Site, Noorderwijk
  - Research Site, Oelegem
  - Research Site, Olen
  - Research Site, Ostend
  - Research Site, Ottignies
  - Research Site, Oudenaarde
  - Research Site, Paal-Beringen
  - Research Site, Paliseul
  - Research Site, Petit-Rechain
  - Research Site, Poederlee
  - Research Site, Pondrôme
  - Research Site, Reet
  - Research Site, Rijkevorsel
  - Research Site, Roeselare
  - Research Site, Ronquière
  - Research Site, Rumbeke
  - Research Site, Sankt Vith
  - Research Site, Seraing
  - Research Site, Sibret
  - Research Site, Sint-Eloois-Winkel
  - Research Site, Sint-Niklaas
  - Research Site, Sint-Ulriks-Kapelle
  - Research site, Souvret
  - Research Site, Steenokkerzeel
  - Research Site, Stekene
  - Research Site, Tavier
  - Research Site, Temse
  - Research Site, Terhagen
  - Research Site, Theux
  - Research Site, Thieusies
  - Research Site, Thuin
  - Research Site, Tielt
  - Research Site, Tienen
  - Research Site, Tilff
  - Research site, Tournai
  - Research Site, Tremelo
  - Research Site, Trois-Ponts
  - Research Site, Turnhout
  - Research Site, Uccle
  - Research Site, Vedrin
  - Research Site, Verviers
  - Research site, Villers-Poterie-Charleroi
  - Research Site, Vilvoorde
  - Research Site, Vissenaken
  - Research Site, Vosselaar
  - Research Site, Waregem
  - Research site, Waremme
  - Research site, Welkenraedt
  - Research Site, Wellin
  - Research Site, Westerlo
  - Research Site, Wetteren
  - Research Site, Wilrijk
  - Research Site, Yvoir
  - Research Site, Zeebrugge
  - Research Site, Zele
  - Research Site, Zemst
  - Research Site, Zoersel
  - Research site, Zottegem
  - Research Site, Zulte
  - Research Site, Zwalm
  - Research Site, Zwevegem
- Luxembourg (4):
  - Research Site, Esch-sur-Alzette
  - Research site, Luxembourg
  - Research Site, Niedercorn
  - Research Site, Warken

REFERENCES:
- [Derived] Louis R, Joos G, Michils A, Vandenhoven G. A comparison of budesonide/formoterol maintenance and reliever therapy vs. conventional best practice in asthma management. Int J Clin Pract. 2009 Oct;63(10):1479-88. doi: 10.1111/j.1742-1241.2009.02185.x. PMID 19769705